CLINICAL TRIAL: NCT03707353
Title: A Phase I/IIa Sporozoite Challenge Study to Assess the Safety, Immunogenicity and Protective Efficacy of Intravenous Boosting With Malaria Vaccine Candidates ChAd63 and MVA Encoding ME-TRAP
Brief Title: An Efficacy Study of IV Boosting With ChAd63/MVA ME-TRAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC066
Record Dates: First submitted 2018-10-10; First posted 2018-10-16 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-07

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1 (Experimental): Volunteers will receive ChAd63 ME-TRAP vaccination intramuscularly, then MVA ME-TRAP vaccination intramuscularly followed by ChAd63 ME-TRAP vaccination intravenously.
  Interventions: Biological: ChAd63 ME-TRAP and MVA ME-TRAP vaccination
- Group 2 (Experimental): Volunteers will receive ChAd63 ME-TRAP vaccination intramuscularly, then MVA ME-TRAP vaccination intramuscularly followed by MVA ME-TRAP vaccination intravenously.
  Interventions: Biological: ChAd63 ME-TRAP and MVA ME-TRAP vaccination
- Group 3 (Experimental): Volunteers will receive ChAd63 ME-TRAP vaccination intramuscularly, followed by ChAd63 ME-TRAP vaccination intravenously.
  Interventions: Biological: ChAd63 ME-TRAP and MVA ME-TRAP vaccination
- Group 4 (Experimental): Volunteers will receive ChAd63 ME-TRAP vaccination intramuscularly, followed by MVA ME-TRAP vaccination intravenously. 4 weeks after the last vaccine dose, all vaccinated volunteers will undergo malaria challenge by mosquito bite.
  Interventions: Biological: ChAd63 ME-TRAP and MVA ME-TRAP vaccination
- Group 5 (No Intervention): 6 Volunteers will receive no vaccinations but will undergo malaria challenge infection by mosquito bite at the same time as groups 1-4.
- Group 6 (No Intervention): 6 Volunteers will be used as infectivity controls if any volunteers from Groups 1-4 are rechallenged 5 - 7 months after the initial CHMI.
- Group A (Experimental): Volunteers will receive ChAd63 ME-TRAP vaccination intramuscularly, then MVA ME-TRAP vaccination intramuscularly followed by MVA ME-TRAP vaccination intravenously.
  Interventions: Biological: ChAd63 ME-TRAP and MVA ME-TRAP vaccination

INTERVENTIONS:
Biological: ChAd63 ME-TRAP and MVA ME-TRAP vaccination — vaccination with ChAd63 ME-TRAP 5x10^10 vp (intramuscularly and intravenously) vaccination with MVA METRAP 2x10^8 pfu (intramuscularly) and MVA METRAP 2x10^7 pfu (intravenously) Group 5 will be challenged with malaria by mosquito bite.
  Arms: Group 1; Group 2; Group 3; Group 4; Group A

SUMMARY:
Plasmodium falciparum Malaria remains a major global health problem with approximately 200 million cases and 500,000 deaths worldwide annually, mostly in African infants. Current malarial control strategies are threatened by emergence of parasite resistance to drug treatment and resistance of the mosquito vector to certain insecticides. A deployable malaria vaccine is therefore a key strategy for reducing malaria mortality and progressing towards global eradication, but those in clinical trials are currently someway short of WHO targets.

ChAd63 ME-TRAP and MVA ME-TRAP are leading candidate vaccines being developed by Adrian Hill's group at the University of Oxford, and collaborators. Since 2007, testing of these vaccines intramuscularly in over 900 volunteers has shown them to be safe, well tolerated and capable of delivering partial efficacy against malaria infection. This study will be the first time studying the efficacy of giving a boosting dose of the vaccines intravenously in what the investigators call a "prime-target" strategy. It follows very encouraging pre-clinical work showing this route can target desirable immune responses to the liver to fight a crucial stage of malaria infection. An ongoing recent phase I study is dose escalating both these vaccines intravenously as a single dose prior to commencing this trial where intramuscular and intravenous doses will be combined for the first time. The investigators will initially recruit 46 healthy UK adult volunteers who will be enrolled into 4 vaccination arms (10 volunteers each) and an unvaccinated control group (6 volunteers) who will undergo a controlled human malaria infection (CHMI). These are standardised, carefully supervised infection experiments used internationally to assess vaccine efficacy. As this is the first time giving intramuscular and intravenous doses of these vaccines in a combined schedule, the investigators will closely profile the safety and immune response during the vaccination follow-up. All trial activity will take place in Oxford.

DETAILED DESCRIPTION:
The study is considered of low risk to the health of participants. Volunteers will receive investigational vaccines, be infected with malaria by mosquito bite, may develop clinical malaria disease, will be treated with antimalarial drugs, and will have blood taken regularly. They will also be given the option to undergo a minimally invasive procedure - Fine Needle Aspiration of the liver - to examine the immune response in this target organ which is also considered to be low risk.

As this is the first time intravenous dose of the vaccines following intramuscular prime/boost doses will be administered, once volunteers have received their intramuscular doses the investigators will stagger the intravenous vaccinations to allow for interim safety reviews. The first volunteer in groups 1&2, once they have received their two intramuscular doses, will receive their intravenous vaccine dose alone and observed for a minimum 8 hours. If there have been no concerns identified at the 8 hour and 24 hour reviews identified by the CI and Local Safety Committee (LSC) chair, the next two volunteers in these groups will receive their intravenous vaccine dose. There will be a further safety 24 hours after these volunteers have been vaccinated before the remaining volunteers are vaccinated.

Volunteers are expected to have both vaccine site reactions (eg, pain, swelling, warmth in the arm where the vaccine is given) and systemic reactions to vaccination (eg, fever, headache, tiredness, sore muscles and joints). These are expected to resolve completely within several days, and symptoms strong enough to prevent usual activities over this time are expected to be uncommon.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent to participate in the trial.
* Agreement to refrain from blood donation during the course of the study and for at least 3 years after the end of their involvement in the study.
* Reachable (24/7) by mobile phone during the period between CHMI and completion of antimalarial treatment.
* Willingness to provide a named person who may be contacted in the event it is not possible to locate the volunteer following CHMI
* Willingness to take a curative anti-malaria regimen following CHMI.
* For volunteers not living in Oxford: agreement to stay in a hotel room close to the trial centre during a part of the study (from at least day 6.5 post mosquito bite until anti-malarial treatment is completed).
* Answer all questions on the informed consent quiz correctly.

Exclusion Criteria:

History of clinical malaria (any species).

* Travel to a clearly malaria endemic locality during the study period or within the preceding six months
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data as assessed by the investigator. This may include non-malaria adenovirus vectored experimental vaccine. If any volunteers undergo rechallenge, this exclusion criterion does not extend to the vaccines previously received in the VAC066 trial.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products, Kathon) or malaria infection.
* Any history of anaphylaxis post vaccination.
* History of clinically significant contact dermatitis.
* Pregnancy, lactation or intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested (described in section 9.6.1).
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Clinically significant disturbances of electrolyte balance, eg, hypokalaemia or hypomagnesaemia
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
* History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait or any haematological condition that could affect susceptibility to malaria infection.
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone.
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone.
* Contraindications to the use of both Riamet and Malarone.
* Any clinical condition known to prolong the QT interval and existing contraindication to the use of Malarone.

Family history of congenital QT prolongation or sudden death and existing contraindication to the use of Malarone.

* History of cardiac arrhythmia, including clinically relevant bradycardia and existing contraindication to the use of Malarone.
* Positive family history in both 1st and 2nd degree relatives < 50 years old for cardiac disease.
* Volunteer unable to be closely followed for social, geographic or psychological reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of intramuscular vaccination followed by intravenous boosting with ChAd63 and MVA encoding ME-TRAP, in healthy malaria-naïve volunteers, assessed by frequency of adverse events | Solicited and Unsolicited AEs will be collected for 28 days. SAEs will be collected from enrolment until the end of the follow-up period (16 weeks following completion of the prime target regimen)
  Occurrence of solicited and unsolicited local and systemic adverse events

SECONDARY OUTCOMES:
To assess cell-mediated immunogenicity generated in malaria naïve individuals of vaccination schedules incorporating intramuscular prime dose(s) followed by intravenous booster with ChAd63 and MVA encoding ME-TRAP. | Up to 11-13 months from initial vaccination
  The key measure of immunogenicity will be ELISPOT to enumerate IFN-γ producing T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V Hill, DPhill FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, UK
Locations (4):
- United Kingdom (4):
  - NIHR Clinical Research Facility, Hammersmith Hospital, London
  - CCVTM, University of Oxford, Oxford
  - John Radcliffe Hospital, Oxford
  - Southampton National Institute for Health Research, Southampton